CLINICAL TRIAL: NCT06981169
Title: PROPULSION SANTE: Inflammometry to Improve the Diagnostic Trajectory in Situations of Suspected Asthma in Children and Adults
Acronym: PROPULSION
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: AstraZeneca (Industry); Niox Group Plc (Unknown); Ministere de la Sante et des Services Sociaux (Other); Association Pulmonaire du Quebec (Other); Fonds recherche du Québec Santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: MP-31-2025-5593
Record Dates: First submitted 2025-04-30; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-02

CONDITIONS: Asthma; Inflammation; Asthma in Children
Keywords: Diagnosis; Asthma; inflammation; FeNO; Blood eosinophil count
MeSH Terms: conditions — Asthma; Inflammation; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, urine, nasal epithelial lining fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged ≥6 years awaiting respiratory function tests requested by primary care: People aged ≥6 years waiting for their respiratory test will be invited to a clinical appointment and offered additional evaluation as part of this study, including : 1/ medical history 2/ exhaled fraction of nitric oxide FeNO measurement (using a portable NIOX VERO device) 3/ a blood test to measure blood eosinophil count (BEC) 4/Questionnaires to be completed on quality of life and asthma control, as well as satisfaction forms.
  Interventions: Diagnostic Test: FeNO; Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: FeNO — FeNO measured with a NIOX VERO device before the respiratory test
Diagnostic Test: blood sample — Blood sample for measuring the blood eosinophil count

SUMMARY:
The objective of this observational study is to assess the relevance of inflammometry (based on the measurement of fractional exhaled nitric oxide (FeNO) and blood eosinophil count (BEC)) as a tool for prioritizing respiratory diagnostic tests.

The study will evaluate the role of inflammometry (FeNO and BEC) in prioritizing diagnostic respiratory tests. It will include patients aged six and older with suspected asthma, referred by non-pulmonologists for diagnostic asthma testing (spirometry or methacholine challenge test) at three hospital centers: Sherbrooke University Hospital Center (CHUS), Sainte-Justine University Hospital Center (CHU Sainte-Justine), and the Montreal Children's Hospital.

The hypothesis is that using inflammometry as a prioritization tool would reduce diagnostic delays for high-risk patients with elevated biomarkers. This study could help shorten wait times, relieve congestion in diagnostic testing queues, and improve the diagnostic pathway. Additionally, it would enhance the interpretation of pulmonary function test results by incorporating inflammometry findings, leading to better patient stratification.

Patients referred from primary care will undergo pulmonary function testing (spirometry ± methacholine challenge) and, as part of the study:

FeNO measurement using a portable device Blood test for eosinophil count Questionnaire on asthma control and quality of life, completed at the visit and at follow-ups at 4, 8, and 12 months

DETAILED DESCRIPTION:
BACKROUND : Asthma is one of the most prevalent chronic diseases worldwide. In Canada, it affects 11% of the population. In Quebec, an estimated 900,000 people suffer from asthma, including 300,000 children. Type 2 eosinophilic inflammation is present in 50% of asthma cases and in 95% of individuals with severe disease, who consume more healthcare resources. This type of inflammation is clinically identified through non-invasive measurements of exhaled nitric oxide (FeNO) and blood eosinophil count (BEC).

Asthmatic patients with Type 2 inflammation are at higher risk of asthma attacks and appear to be at risk of accelerated lung function decline, both in adults and children. The presence of Type 2 inflammation predicts a strong response to inhaled corticosteroids (ICS).

Currently, post-bronchodilator reversibility and/or bronchial hyperresponsiveness documented via spirometry are the two main approved methods for diagnosing asthma. Bronchial provocation testing is required in 80% of suspected asthma cases, but our population faces a severe lack of access to this test.The average wait time for this 1-2 hour procedure exceeds one year in our three centers.

Currently, prioritization is based on the order in which requests are received, with internal referrals given priority over external ones. In Europe, FeNO is already used as a complementary diagnostic tool in primary care, while in Quebec, it is only accessible in severe asthma clinics.

Type 2 eosinophilic inflammation is present in 50% of asthma cases and in 95% of severe asthma cases. This inflammation can be identified through non-invasive biomarkers, such as FeNO and blood eosinophil count. Individuals with type 2 inflammation are at higher risk for asthma attacks and are more likely to experience accelerated decline in respiratory function, both in adults and children. However, type 2 inflammation also predicts a strong response to inhaled corticosteroids (ICS).The identification of these markers represents a treatable trait.

HYPOTHESIS

As a prognostic procedure that identifies a treatable trait, early measurement of inflammatory biomarkers could:

1. Prioritize highly inflamed patients for bronchial provocation testing.
2. Provide personalized therapy based on the inflammation type, with evidence-based recommendations included in the medical reports.
3. Improve the management of asthmatic patients who do not respond to initial treatment, ensuring better access to specialized care.

OBJECTIVES

For patients ≥6 years old with suspected asthma, referred by non-pulmonologists for diagnostic testing, the study aims to use inflammometry to:

1. Reduce diagnostic delays for high-risk patients with probable asthma and exacerbation risk.
2. Enhance test result interpretation by incorporating inflammometry findings, asthma probability assessment, exacerbation risk, and expected response to anti-inflammatory therapies.
3. Alleviate waiting lists across our three centers.
4. Analyze and optimize the diagnostic pathway for suspected asthma cases in Quebec by generating real-world evidence on the clinical, economic, and environmental benefits of inflammometry.

METHODOLOGY For one year, an additional respiratory therapist at each center will conduct diagnostic tests for suspected asthma (spirometry with pre/post-bronchodilator testing or methacholine challenge) requested by non-pulmonologists at the Sherbrooke University Hospital Center (CHUS), CHU Sainte-Justine, and the Montreal Children's Hospital.

All patients ≥6 years old on the waiting list will be invited to a clinic visit, where a complementary assessment will be offered. This innovative approach includes:

1. FeNO measurement (exhaled air)
2. Blood eosinophil count (capillary or venous sample)
3. Questionnaires on asthma control and quality of life, completed at baseline and at 4, 8, and 12 months

If spirometry is non-diagnostic, bronchial provocation will be prioritized based on inflammatory profile:

1. if ≥1 biomarker is elevated (for those ≥12 years old, FeNO ≥25 ppb or blood eosinophils ≥300 cells/µL; for those aged 6-<12 years, FeNO ≥20 ppb or eosinophils ≥300 cells/µL), the bronchial provocation test will be prioritized (<2-4 weeks).
2. If both biomarkers are low, the scheduling of the provocation test will follow the usual timelines.

If spirometry or provocation confirms asthma, additional biomarker data will inform the physician about the risk of asthma attacks.

OUTCOMES The primary outcome will be diagnostic delay evolution for high- vs. low-risk asthma patients, analyzed before, during, and after the project.

Receiver Operating Characteristic (ROC) curves will be used to assess the diagnostic performance of inflammometry as a potential diagnostic tool, including determining thresholds that could eliminate the need for provocation test. The analyses will be completed by questionnaires evaluating user satisfaction, economic efficiency measures (cost-effectiveness, cost-utility, budget impact), and an environmental impact assessment (measured in kgCO2 emitted by inhalers used when asthma is not diagnosed).

IMPACT

1/ Implementation of an evidence-based prioritization system for primary care referrals, substituting the current chronological approach, to reduce wait times for high-risk patients. 2/ Integrating biomarker results with pulmonary function test outcomes will refine their interpretation and better assess the likelihood of an asthma diagnosis, exacerbation risk, and response to anti-inflammatory treatments. 3/The resources allocated by this project will help reduce waitlists. 4/ Real-world evidence from Quebec will be used to improve the asthma diagnostic algorithm, facilitating the integration of inflammometry into asthma diagnosis in the province. This could potentially eliminate 20% of bronchial provocation tests, reducing costs with net-zero financial impact.

ELIGIBILITY:
Inclusion Criteria:

* patients age 6 and older
* referred by primary care ofr an asthma diagnostic test (spirometry or methacholine challenge)

Exclusion Criteria:

* referred by pulmonologist

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with asthma-suggestive symptoms, referred to Sherbrooke Universty Hospital Center (CHU), CHU Sainte-Justine, and the Montreal Children's Hospital by a non-pulmonologist healthcare professional for asthma diagnosis (pre/post-bronchodilator spirometry and, if non-diagnostic, a methacholine bronchial provocation), will be scheduled for an appointment with the project's designated respiratory therapist .
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the diagnostic delay for asthma in patients with high risk due to elevated inflammatory markers versus those with low risk | At the time of the methacholine challenge test
  The average delay before the implementation of the project will be calculated based on 25 methacholine challenge tests requested by primary care and performed before the project.The average time during implementation will be analyzed continuously, both overall and in subgroups based on inflammatory status.

SECONDARY OUTCOMES:
Impact of inflammatory status on quality of life according astshma control before and after diagnostic testing | at the baseline, then 4, 8, 12 month
  Comparison of Asthma Control Questionnaire
Diagnostic performance of fractional exhaled nitric oxide (FeNO) | At the time of the methacholine challenge test
  ROC curve analysis of FeNO values. The diagnosis of asthma will be confirmed by a positive methacholine challenge with a dose provocation (DP20) <400 mcg (equivalent of concentration provocation (CP20) <16 mg/mL). An exploratory analysis following European standards (DP20 ≤ 200 mcg or CP20 ≤ 8 mg/mL28-30) will also be conducted.
Diagnostic performance of Blood eosinophils count | At the time of the methacholine challenge test
  ROC curve analysis of BEC values. The diagnosis of asthma will be confirmed by a positive methacholine challenge with a DP20 <400 mcg (CP20 <16 mg/mL). An exploratory analysis following European standards (DP20 ≤ 200 mcg or CP20 ≤ 8 mg/mL28-30) will also be conducted.
Comparison of the Economic Efficiency of Asthma Diagnostic Algorithms | baseline visit up to 12 months after the diagnostic tests
  Sum of health expenses attributable to asthma for the participant in Canadian dollar, including medication, hospitalization, estimation
Analysis of user satisfaction questionnary regarding inflammometry | baseline visit
  Qualitative descriptive analysis of user satisfaction questionnary regarding inflammometry. Responses will be analyzed by group (patients, legal guardian) and based on whether an asthma diagnosis was confirmed or not.4 questions (inflammatory assessment, blood test, respiratory test, long wait for diagnostic test) on 5-level sides (strongly agree, agree, neutral, disagree, strongly disagree)
Evaluation of the environmental impact | baseline visit up to 12 months after the diagnostics tests
  Estimation of the carbon footprint (in kgCO2) of the asthma diagnostic delay. This estimation will be limited to calculating the annualized CO2 burden of inhalers dispensed to non-asthmatic individuals awaiting their diagnostic tests. The carbon footprint per inhaler will be sourced from Cascades Canada
Evaluation of asthma control according to medication use | At the time of the initial visit, then at the 4, 8 and 12-month follow-up questionnaires
  Comparison of asthma medication consumption before and after diagnosis, including number of inhalers, and initiation or change of treatment, by querying the dossier santé québec and then by questionnaire sent during virtual follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data of this study may be shared if the investigators proposed use of the data has been approved by the study principal investigator and an institutional research ethics committee.
Time Frame: up to 2035
Access Criteria: Data of this study may be shared if the investigators proposed use of the data has been approved by the study principal investigator and an institutional research ethics committee.

REFERENCES:
- [Derived] Gronnier M, Desy L, Pouliot L, Lemieux SE, Vezina FA, Lachapelle P, Counil FP, Duval M, Cliche D, Lemaire-Paquette S, Coulibaly L, Hudon C, Lands LC, Ducharme FM, Tse S, Couillard S. Integrating blood eosinophils and exhaled nitric oxide (FeNO) in asthma diagnostic pathways for adults and children: the PROPULSION SANTE observational study with translational sub-studies (DIVE, DIVE2)-protocols. BMJ Open Respir Res. 2025 Nov 27;12(1):e003750. doi: 10.1136/bmjresp-2025-003750. PMID 41314665